CLINICAL TRIAL: NCT06518291
Title: COMPARISON OF NITROFURANTOIN WITH FOSFOMYCIN in TREATING CYSTITIS IN WOMEN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shalamar Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sheema Yousuf, Doctor, Shalamar Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-741
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Nitrofurantoin; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- nitrofurantoin group (Active Comparator)
  Interventions: Drug: Nitrofurantoin 100 MG
- Fosfomycin group (Active Comparator)
  Interventions: Drug: Fosfomycin

INTERVENTIONS:
Drug: Nitrofurantoin 100 MG — Comparing two drugs in UTI treatment
  Arms: nitrofurantoin group
Drug: Fosfomycin — treatment of UTI
  Arms: Fosfomycin group

SUMMARY:
Fosfomycin and nitrofurantoin are increasingly being prescribed in outpatients for the oral treatment of urinary tract infection (UTI). The newest guidelines for empirical treatment of women with uncomplicated urinary tract infections (UTIs) advise clinicians to choose among three venerable antibiotics: trimethoprim-sulfamethoxazole, nitrofurantoin, and fosfomycin. Although both nitrofurantoin and fosfomycin have shown efficacy against most urinary pathogens, no recent head-to-head comparisons have been reported. So, this study will be conducted to compare effectiveness of both drugs.

DETAILED DESCRIPTION:
INTRODUCTION Urinary tract infection (UTI) is a broad term that encompasses a spectrum of infectious syndromes that affect the urinary tract anywhere from the urethra to the kidneys. UTIs are one of the most common infections, and it is reported that 50%-60% of women have at least one UTI in their lifetime.1 It is the second most common reason for antibiotic prescriptions, after respiratory tract infections.2 Acute uncomplicated cystitis is an infection of the bladder and urethra that affects mainly women and girls from 2 years of age and pyelonephritis is an infection of the renal parenchyma. Escherichia coli is the most common causative pathogen of both diseases and accounts for approximately 85% of community-acquired UTIs and 50% of hospital-acquired UTIs.3,4,5 There have been recent reports of an increasing level of antibiotic resistance in pathogens causing uncomplicated UTIs.6,7 The 2017-2018 WHO GLASS (Global Antimicrobial Resistance and Use Surveillance System) report indicates >70% resistance to ceftriaxone and ciprofloxacin in E. coli isolated from UTIs in Pakistan.7,8 A previous study on UTI pathogens in Karachi found that 49% of Gram-positive and 57% of Gram-negative bacteria were resistant to ciprofloxacin.5,9 Despite of this, ciprofloxacin is readily available over the counter in an oral suspension throughout Pakistan and is prescribed widely by physicians.9 This high level of resistance indicates that the use of the antibiotic as a first-line treatment for UTI in Pakistan needs to be reconsidered. It has been shown in studies that there is low resistance rates to fosfomycin and nitrofurantoin.10,11,12,13,14 Given increasing antimicrobial resistance, guidelines for the treatment of uncomplicated lower urinary tract infections (UTIs) were modified in 2010 to recommend nitrofurantoin and fosfomycin as first-line agents; their use has since increased exponentially.3,12,15Worldwide first-line agents for uncomplicated UTIs include nitrofurantoin, sulfamethoxazole/trimethoprim and fosfomycin.16 Nitrofurantoin is bacteriostatic, not bactericidal, and must be used for 5 to 7 days. It is the preferred drug for low-dose long-term prophylaxis in patients with recurrent UTIs.17 Fosfomycin is FDA-approved as a 3gram single-dose therapy for uncomplicated UTIs.18 A single dose will provide therapeutic urinary concentrations for 2 to 4 days and is comparable to 7- to 10-day therapy with other agents.18,19

OBJECTIVE As the use of nitrofurantoin and fosfomycin has increased since guidelines began recommending them as first-line therapy for lower urinary tract infection (UTI). This study will be conducted to compare the clinical and microbiologic efficacy of nitrofurantoin and fosfomycin in women with cystitis.

RATIONALE Fosfomycin and nitrofurantoin are increasingly being prescribed in outpatients for the oral treatment of urinary tract infection (UTI). The newest guidelines for empirical treatment of women with uncomplicated urinary tract infections (UTIs) advise clinicians to choose among three venerable antibiotics: trimethoprim-sulfamethoxazole, nitrofurantoin, and fosfomycin. Although both nitrofurantoin and fosfomycin have shown efficacy against most urinary pathogens, no recent head-to-head comparisons have been reported. So, this study will be conducted to compare effectiveness of both drugs.

OPERATIONAL DEFINITIONS:

1. Cystitis is infection of urinary bladder. Uncomplicated cystitis refers to lower urinary tract infection in women who are otherwise healthy. Complicated cystitis is associated with risk factors (diabetes, renal transplantation, pregnancy, immunocompromised, indwelling catheter, abnormality of urinary tract) that increase the chances of antibiotic failure.20
2. Pyelonephritis is infection of renal parenchyma resulting in fever, pain in lumber region and vomiting.
3. Adverse effects of Nitrofurantoin: Headache, dizziness, nausea, diarrhea, vomiting, loss of appetite, chest pain, numbness in hands and feet, brown urine.20
4. Adverse effects of Fosfomycin: vaginal discharge, abdominal pain, headache, back pain, bodyaches , indigestion, dryness of throat, heavy painful menstruation, skin rash, weakness.20
5. Clinical response was defined as clinical resolution (complete resolution of symptoms and signs of urinary tract infection without prior failure).
6. Clinical failure (need for additional or change in, antibiotic treatment due to a urinary tract infection, or discontinuation due to lack of efficacy).
7. Indeterminate (either persistence of symptoms without objective evidence of infection or any extenuating circumstances precluding a classification of clinical resolution/failure).
8. Microbiologic response was defined as resolution (eradication of the infecting strain with no recurrence of bacteriuria [<103 colony-forming units/mL] during follow-up) or failure (bacteriuria ≥103 colony- forming units/mL with the infecting strain).21

METHODOLOGY Study Design: Randomized clinical trial Sampling Technique: Simple random sampling Study duration: six months Settings: Outpatient Gynae Department Shalamar Hospital Lahore

Study will be conducted after IRB approval.

Sample Size Calculation

Given:

Effectiveness of Drug 1, nitrofurantoin(p1) = 90% =0.90 22,23 Effectiveness of Drug 2, fosfomycin(p2) =80%=0.80 22,23 Significance level (α)=0.05 Power (1-β) =0.80

The sample size (n) for each group can be calculated using the following formula:

n= (Z α/2 +Z β)2 x {p1(1- p1) + p2(1- p2)}/ (p1- p2)2

where:

Z α/2 is the critical value from the standard normal distribution for a tow tailed test at significance level α. For α=0.05, Z α/2 =1.96.

Z β is the critical value from the standard normal distribution for the desired power. For a power of 0.80, Z β =0.84

Calculating the combined variance:

p1(1- p1) =0.90x0.10+0.09 p2(1- p2) =0.80x0.20=0.16 p1(1- p1) + p2(1- p2) = 0.09+0.16=0.25

Calculating the squared difference in proportions:

(p1- p2)2 = (0.90-0.80)2 =0.102 =0.01

Putting the values in the formula:

n= {(1.96+0.84)2x0.25}/ 0.01= 1.96/0.01=196 Each group requires 196 patients, making the total sample size of 392

Intervention and Procedures Participants will be randomly assigned to either oral Nitrofurantoin 100 mg 3 times a day for 5 days or a single 3-g dose of oral Fosfomycin and instructed to contact study investigators in the absence of clinical improvement. They will attend follow-up visits at 7 and 14 days after completion of antibiotic therapy. Urine cultures will be collected before starting antibiotic. Because of fosfomycin's long half-life,24 antibiotic therapy will be considered completed in both groups on day 5 after randomization.

Voided midstream urine specimens will be collected in sterile containers and transported within 24 hours to laboratory, where specimens will be cultured according to published recommendations. Cultures will be reported positive when 103 cfu/mL or more of at least 1 bacterium was detected.20

Data Analysis

Analysis will be performed by using SPSS version 21. Baseline characteristics will be described by mean and standard deviation. The clinical and bacteriologic resolution will be compared between treatment groups using the Chi square test; incidence of adverse events and other outcome measures will be compared using the Fisher exact test. Patients who will show documented clinical failure and were then lost to follow-up will be included in the primary outcome analysis of any failure by day 14, while those whose response status was unknown before dropout were considered missing; missing values were excluded from the primary analysis. P value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged 18 years and older presenting with at least 1 symptom of lower UTI such as dysuria, urgency, frequency, or suprapubic tenderness and a urine dipstick test result positive for either nitrites or leukocyte esterase. Confirmed UTI will require the presence of at least 1 of the 4 urinary symptoms required for inclusion and a positive urine culture (≥103 cfu/mL). 21

Exclusion Criteria:

* 1) Pregnancy and lactation 2) Suspected upper UTI (presence of fever, chills, or flank pain) 3) Antibiotic use or any symptoms consistent with UTI in the preceding 4 weeks 4) Indwelling urinary catheter or otherwise complicated UTI 5) Immunosuppression (untreated infection with HIV, ongoing chemotherapy or radiation therapy, use of high-dose corticosteroids or other immunosuppressive medication) 6) Renal insufficiency (creatinine clearance <30 mL/min).

Ages: 18 Years to 83 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
clinical response following completion of therapy by history | 7 days

SECONDARY OUTCOMES:
bacteriologic response after therapy completion by urine culture test result | 14 days

IPD SHARING:
Plan to Share IPD: No